CLINICAL TRIAL: NCT01433081
Title: The Effect of Magnesium Sulfate Infusion on the Quality of Recovery of Ambulatory Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Gildasio De Oliveira, Gildasio De Oliveira, M.D. Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STU00032878
Record Dates: First submitted 2011-09-09; First posted 2011-09-13 (Estimated); Results first posted 2014-04-02 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-02

CONDITIONS: Pain; Opioid Use, Unspecified, Uncomplicated
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnesium sulfate infusion (Active Comparator): Administration of magnesium suflate
  Interventions: Drug: administration of magnesium sulfate
- Placebo (Placebo Comparator): .9 normal saline infusion
  Interventions: Drug: Placebo infusion of .9 normal saline

INTERVENTIONS:
Drug: Placebo infusion of .9 normal saline — administration of .9 normal saline
  Arms: Placebo
Drug: administration of magnesium sulfate — administration of magnesium sulfate
  Arms: Magnesium sulfate infusion

SUMMARY:
A national survey has revealed that 80% of patients experienced pain after surgery and 86% of these patients had moderate, severe or extreme pain (1).Postoperative pain can extend recovery room stay after surgery and it is also a common cause of unanticipated admissions which have important economic implications(2).More importantly, postoperative pain can lead to a poor quality of recovery in ambulatory patients. The Intraoperative use of medications that might decrease postoperative pain is therefore highly desirable.

Some medications such as lidocaine and ketamine have been proved to decrease postoperative pain when given during the Intraoperative period in ambulatory patients(3,4) but it is still unknown if those medications can in fact lead to a better quality of recovery .

Magnesium sulfate is a non-competitive calcium antagonist at the N-methyl-D- aspartate (NMDA) receptor(5). NMDA receptors have an important role on pain modulation (6). The use of Intraoperative magnesium in order to decrease postoperative pain had contradictory results in different studies. Some studies have shown a potential benefit of magnesium in decreasing postoperative pain (7,8) while others have not demonstrated any benefit (9,10).

In the ambulatory setting, specifically, Tramer et al. did not find any improvement on postoperative pain after an Intraoperative dose of magnesium for patients undergoing ilioinguinal hernia repair(11). Koinig et al., however, demonstrated a significant reduction in the postoperative analgesic requirements in patients undergoing arthroscopic knee surgery (12).

Even though, the reduction of postoperative opioid requirement has been used in many studies in the ambulatory literature, it has been recently questioned by some investigators (13).Patients might take more opioid medications but they may not necessarily develop opioid related side effects such as nausea and vomiting. A more global evaluation of the patient involving several aspects of recovery would be more significant.

The modified quality of recovery 40(MQOR40) is a validated 40 item instrument to assess the quality of postoperative recovery (14). Myles et al. concluded that the MQOR40 would be a useful outcome measure to assess the impact on changes in health care delivery (15), but anesthesia studies underutilize this instrument.

As more complex and painful procedures are being done in the ambulatory setting , the use of non-opioid strategies to control postoperative pain and to enhance quality of recovery will have even a greater role in the anesthetic management of patients. Magnesium has not been established as a potential adjuvant in ambulatory patients with conflicting results of previous investigators. The main objective of this study is to evaluate if the Intraoperative use of magnesium have the ability to improve postoperative quality of recovery in ambulatory patients.

ELIGIBILITY:
Inclusion Criteria:

* undergoing lumpectomy
* ASA I and II
* Age between 18-64

Exclusion Criteria:

* pregnancy
* breastfeeding -history of EKG abnormalities-
* kidney disease including: End Stage Renal Disease and polycystic kidney disease
* unable to understand the informed consent
* use of opioid in the last week
* use of calcium channel blockers
* Drop-out: surgeon or patient request

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gildasio De Oliveira, MD, Principal Investigator — Northwestern University
Locations (1):
- Prentice Womens Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Apfelbaum JL, Chen C, Mehta SS, Gan TJ. Postoperative pain experience: results from a national survey suggest postoperative pain continues to be undermanaged. Anesth Analg. 2003 Aug;97(2):534-540. doi: 10.1213/01.ANE.0000068822.10113.9E. PMID 12873949
- [Background] White PF. Multimodal analgesia: its role in preventing postoperative pain. Curr Opin Investig Drugs. 2008 Jan;9(1):76-82. PMID 18183534
- [Background] McKay A, Gottschalk A, Ploppa A, Durieux ME, Groves DS. Systemic lidocaine decreased the perioperative opioid analgesic requirements but failed to reduce discharge time after ambulatory surgery. Anesth Analg. 2009 Dec;109(6):1805-8. doi: 10.1213/ANE.0b013e3181be371b. PMID 19923506
- [Background] Berti M, Baciarello M, Troglio R, Fanelli G. Clinical uses of low-dose ketamine in patients undergoing surgery. Curr Drug Targets. 2009 Aug;10(8):707-15. doi: 10.2174/138945009788982496. PMID 19702519
- [Background] Mayer ML, Westbrook GL, Guthrie PB. Voltage-dependent block by Mg2+ of NMDA responses in spinal cord neurones. Nature. 1984 May 17-23;309(5965):261-3. doi: 10.1038/309261a0. PMID 6325946
- [Background] Begon S, Pickering G, Eschalier A, Mazur A, Rayssiguier Y, Dubray C. Role of spinal NMDA receptors, protein kinase C and nitric oxide synthase in the hyperalgesia induced by magnesium deficiency in rats. Br J Pharmacol. 2001 Nov;134(6):1227-36. doi: 10.1038/sj.bjp.0704354. PMID 11704642
- [Background] Ryu JH, Kang MH, Park KS, Do SH. Effects of magnesium sulphate on intraoperative anaesthetic requirements and postoperative analgesia in gynaecology patients receiving total intravenous anaesthesia. Br J Anaesth. 2008 Mar;100(3):397-403. doi: 10.1093/bja/aem407. PMID 18276652

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled consecutively from 2/2011 through 4/2013.
Groups:
- Placebo: Normal saline infusion
Period: Overall Study
Arm/Group | Magnesium Sulfate Infusion | Placebo
Started | 25 | 25
Completed | 23 | 23
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Magnesium Sulfate Infusion | Placebo | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (6.15) | 52 (7.7) | 52 (7.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Quality of Recovery Scores Post Operative
Description: Quality of recovery scores post operative. Scored on a scale of 40 (poor recovery) to 200 (good recovery).
Time Frame: 24 hours post operative
Population: Two drop outs for either arm were removed from analysis.
Measure: Mean (Inter-Quartile Range); unit: units on scale 40 (low) - 200 (high)
Arm/Group | Magnesium Sulfate Infusion | Placebo
Number analyzed (Participants) | 23 | 23
units on scale 40 (low) - 200 (high) | 183 [173 to 188] | 159 [153 to 175]

2. Secondary Outcome: Opioid Consumption
Description: Opioid consumption after discharge
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: miligram morphine equivalents
Arm/Group | Magnesium Sulfate Infusion | Placebo
Number analyzed (Participants) | 23 | 23
miligram morphine equivalents | 10 [0 to 20] | 30 [20 to 40]

ADVERSE EVENTS:
Time Frame: 24 hours
Description: Nausea in the post operative period
Arm/Group | Magnesium Sulfate Infusion | Placebo
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 7/23 | 10/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Magnesium Sulfate Infusion (N=23) | Placebo (N=23)
Nausea (Gastrointestinal disorders) | 7 (10) | 10 (10) — Nausea in 24 hour post operative period.
Vomiting (Gastrointestinal disorders) | 2 (2) | 6 (6) — Vomiting in 24 hour period post operative.

LIMITATIONS AND CAVEATS:
We only examined subjects with normal kidney function that were at low risk for magnesium toxicity. It is possible that the current intervention regimen could have led to toxic levels in higher risk patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No